CLINICAL TRIAL: NCT02521558
Title: Effectiveness of Home-based Electronic Cognitive Therapy in Alzheimer's Disease
Acronym: CTAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was halted early because of low adherence to the intervention.
Sponsor: Boston University (Other)
Collaborators: Wallace H. Coulter Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-34203
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Memory Disorders; Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Cognitive rehabilitation; Mobile electronic application; Memory tasks
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction; Alzheimer Disease | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the Intervention Group, patients will receive an iPad with the Constant Therapy cognitive rehabilitation application. Patients in the Intervention Group will practice the memory tasks developed for the Constant Therapy application for a total of six months. On a weekly basis, a clinician and/or research assistant will check in with the patient to answer any questions or address any concerns the patient has with using the Constant Therapy application, or how to perform any of the memory tasks. At the end of six months, each individual in the Intervention Group is assessed with standard cognitive testing to determine if there was any change on overall cognition.
  Interventions: Behavioral: Intervention Group
- Control Group (Active Comparator): The Control Group will not receive any intervention. The Control Group will be given simple sets of puzzle booklets to practice over the 6 month period (e.g., word search puzzles, number and/or math puzzles). The Control Group will also receive standardized cognitive testing at the end of 6 months. Weekly check-ins by a clinician and/or research assistant will also occur in the Control Group. Every 4th patient recruited for the study will be assigned to the Control Group.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Intervention Group — The investigators are interested in how practicing memory tasks can improve memory in patients with MCI and with AD. Specifically, patients will perform a set of cognitive rehabilitation tasks designed to train memory in order to determine if these tasks are effective in improving memory or slowing the progression of Alzheimer's disease. Patients will practice memory tasks for about an hour daily, for a total duration of 6 months. A research assistant or clinician will conduct weekly check-ins with each participant assess whether or not participants in the Intervention Group exhibit weekly improvements and to determine if patients are regularly adhering to the tasks.
  Arms: Intervention Group
Behavioral: Control Group — The Control Group will not receive any cognitive rehabilitation tasks for a six month period. Instead, they will simply be given booklets of puzzles (e.g., word search, number puzzles, etc.) to work on for the duration of 6 months.
  A research assistant or clinician will conduct weekly check-ins with each participant assess whether or not participants in the control group feel like they are benefiting from the puzzles.
  Participants in the Control Group will be given a standard battery of neuropsychological tests prior to the the puzzles and after the puzzles to assess any changes in memory, language, attention, and executive functioning.
  Arms: Control Group

SUMMARY:
The current study will examine the use of a mobile electronic application used to deliver cognitive rehabilitation to patients with mild cognitive impairment due (MCI) due to Alzheimer's disease (AD), and patients with mild AD. Patients will be given a specific cognitive rehabilitation program on their mobile device (iPad) with specific tasks for them to complete. The goal of this study is to determine if a) patients are able to use and adhere to a cognitive rehabilitation program delivered to their mobile device and b) to determine if patients can improve their language, attention, and memory by completing cognitive rehabilitation tasks assigned to them.

DETAILED DESCRIPTION:
In the current study, the investigators are examining the use of a mobile electronic application used to deliver cognitive rehabilitation tasks to patients with mild cognitive impairment due to Alzheimer's disease, and patients with mild Alzheimer's disease. An estimated 100 patients will be enrolled into the study (~50 patients with mild cognitive impairment, ~50 patients with Alzheimer's disease).

Participants will either receive memory tasks designed to help stabilize or improve memory (Intervention Group) or a set of word or math puzzles (Control Group). Participants will complete memory tasks or puzzles for a six month period. The investigators will conduct pre- and post- neuropsychological testing to assess changes in cognitive status (e.g., memory, language, executive functioning) in the intervention group. Neuropsychological tests assessing changes to cognition will be completed prior to participant assignment to the Intervention or Control Group. Both groups will then be assessed again using neuropsychological tests. The investigators will also assess changes in performance on cognitive rehabilitation tests over the six month period to determine the efficacy of these tasks.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of mild cognitive impairment due to Alzheimer's disease (MCI due to AD) by the patient's referring clinician per recent National Institutes of Aging-Alzheimer's Association criteria (Albert et al., 2011).
* A diagnosis of mild Alzheimer's disease by the patient's referring clinician per recent National Institutes of Aging-Alzheimer's Association criteria (McKhann et al., 2011).
* 50-90 years of age.

Exclusion Criteria:

* Younger than the age of 50 or older than the age of 90.
* Any self-reported history of substance abuse or alcohol abuse.
* Any self-reported history of prior head trauma (e.g., stroke, traumatic brain injury)
* Any prior self-reported history of significant depression or other mood disorder.

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in cognition as measured by the Mini Mental Status Exam | Month 0 (Prior to administration of cognitive rehabilitation tasks) and Month 6 (after administration of cognitive rehabilitation tasks)
  Participants will be administered the Mini Mental Status Exam (MMSE) to both the intervention and control groups. This will occur prior to any to type of intervention (Month 0). Scores on the MMSE range from 0 to 30.
  Specifically the investigators are examining if cognitive status changes as measured by the MMSE prior to intervention (Month 0), and post-intervention (Month 6). The investigators will compare changes in MMSE scores both pre- and post- in the intervention group, but also compare performance on these measures to the control group.
Changes in cognition as measured by the Montreal Cognitive Assessment | Month 0 (Prior to administration of cognitive rehabilitation tasks) and Month 6 (after administration of cognitive rehabilitation tasks)
  Participants will be administered the Montreal Cognitive Assessment (MoCA) to both the intervention and control groups. This will occur prior to any to type of intervention (Month 0). Scores on the MoCA range from 0 to 30.
  Specifically the investigators are examining if cognitive status changes as measured by the MoCA prior to intervention (Month 0), and post-intervention (Month 6). The investigators will compare changes in MoCA scores both pre- and post- in the intervention group, but also compare performance on these measures to the control group.
Changes in cognition as measured by the Consortium to Establish a Registry in Alzheimer's disease Word List Test | Month 0 (Prior to administration of cognitive rehabilitation tasks) and Month 6 (after administration of cognitive rehabilitation tasks)
  Participants will be administered the Consortium to Establish a Registry in Alzheimer's disease Word List Learning Test (CERAD) to both the intervention and control groups. This will occur prior to any to type of intervention (Month 0). The CERAD measures the immediate recall of a list of words (up to 30 correct recall on 3 individual recall trials), delayed recall (up to 10 correct recall after a 5 minute delay), and on yes-no recognition memory (up to 10 correct recognition).
  Specifically the investigators are examining if list learning changes as measured by the CERAD prior to intervention (Month 0), and post-intervention (Month 6). The investigators will compare changes in CERAD scores both pre- and post- in the intervention group, but also compare performance on these measures to the control group.
Changes in cognition as measured Letter and Category Fluency | Month 0 (Prior to administration of cognitive rehabilitation tasks) and Month 6 (after administration of cognitive rehabilitation tasks)
  Participants will be administered the Letter and Category Fluency to both the intervention and control groups. This will occur prior to any to type of intervention (Month 0). For letter fluency, participants name as many words as possible in a minute that start with the letters F, A, and S. For category fluency, participants name as many words as possible in a minute that are within the Animals, Vegetables, and Fruits categories.
  Specifically the investigators are examining if fluency changes as measured by the fluency prior to intervention (Month 0), and post-intervention (Month 6). The investigators will compare changes in fluency scores both pre- and post- in the intervention group, but also compare performance on these measures to the control group.
Changes in cognition as measured by the Boston Naming Test (Short Form) | Month 0 (Prior to administration of cognitive rehabilitation tasks) and Month 6 (after administration of cognitive rehabilitation tasks)
  Participants will be administered the Boston Naming Testing Short Form (BNT-15) to both the intervention and control groups. This will occur prior to any to type of intervention (Month 0). The BNT-15 consists of 15 line drawings (with a maximum score of 15 correct).
  Specifically the investigators are examining if confrontation naming of line drawings as measured by the BNT-15 prior to intervention (Month 0), and post-intervention (Month 6). The investigators will compare changes in fluency scores both pre- and post- in the intervention group, but also compare performance on these measures to the control group.
Changes in cognition as measured by the Trail Making Parts A & B | Month 0 (Prior to administration of cognitive rehabilitation tasks) and Month 6 (after administration of cognitive rehabilitation tasks)
  Participants will be administered the Trail Making Test (Parts A & B) to both the intervention and control groups. This will occur prior to any to type of intervention (Month 0). The Trail Making Test Part A consists of connecting a series a numbers with a line in ascending order as quickly as possible (performance is timed, the score is the time it takes to finish). The Trail Making Test Part B consists of connect a series of letters and numbers, alternating back and forth between them, as quickly as possible in ascending order (performance is timed, the score is the time it takes to finish).
  Specifically the investigators are examining if Trail Making performance as measured by the Trail Making Tests prior to intervention (Month 0), and post-intervention (Month 6). The investigators will compare changes in fluency scores both pre- and post- in the intervention group, but also compare performance on these measures to the control group.

SECONDARY OUTCOMES:
Changes in performance on cognitive rehabilitation tasks (composite measure of memory tasks) | During intervention (6 month time frame, composite measure)
  In the intervention group, the investigators will examine speed and accuracy data on all cognitive rehabilitation memory tasks. Tasks will be converted into a single memory composite measure (for both speed and accuracy data).
  The investigators will cull performance on the tasks on a weekly basis. Weekly data will be treated as a single data points. Participants will be followed for approximately 24 weeks (or 6 months).
  The investigators will use a regression analysis to analyze to determine changes in the slope on speed and accuracy for each of these data points. Additionally, the investigators will use inferential statistics, such as ANOVA, to determine if participants improve on a week by week basis. These analyses will be conducted on the composite of memory data collected from all the memory tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Budson, MD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu F, Rose KM, Burgener SC, Cunningham C, Buettner LL, Beattie E, Bossen AL, Buckwalter KC, Fick DM, Fitzsimmons S, Kolanowski A, Janet K, Specht P, Richeson NE, Testad I, McKenzie SE. Cognitive training for early-stage Alzheimer's disease and dementia. J Gerontol Nurs. 2009 Mar;35(3):23-9. doi: 10.3928/00989134-20090301-10. PMID 19326826
- [Background] Talassi E, Guerreschi M, Feriani M, Fedi V, Bianchetti A, Trabucchi M. Effectiveness of a cognitive rehabilitation program in mild dementia (MD) and mild cognitive impairment (MCI): a case control study. Arch Gerontol Geriatr. 2007;44 Suppl 1:391-9. doi: 10.1016/j.archger.2007.01.055. PMID 17317481
- [Background] Olazaran J, Muniz R, Reisberg B, Pena-Casanova J, del Ser T, Cruz-Jentoft AJ, Serrano P, Navarro E, Garcia de la Rocha ML, Frank A, Galiano M, Fernandez-Bullido Y, Serra JA, Gonzalez-Salvador MT, Sevilla C. Benefits of cognitive-motor intervention in MCI and mild to moderate Alzheimer disease. Neurology. 2004 Dec 28;63(12):2348-53. doi: 10.1212/01.wnl.0000147478.03911.28. PMID 15623698
- [Background] Spector A, Orrell M, Woods B. Cognitive Stimulation Therapy (CST): effects on different areas of cognitive function for people with dementia. Int J Geriatr Psychiatry. 2010 Dec;25(12):1253-8. doi: 10.1002/gps.2464. PMID 20069533
- [Background] Spector A, Thorgrimsen L, Woods B, Royan L, Davies S, Butterworth M, Orrell M. Efficacy of an evidence-based cognitive stimulation therapy programme for people with dementia: randomised controlled trial. Br J Psychiatry. 2003 Sep;183:248-54. doi: 10.1192/bjp.183.3.248. PMID 12948999
- [Background] Burgener SC, Buettner LL, Beattie E, Rose KM. Effectiveness of community-based, nonpharmacological interventions for early-stage dementia: conclusions and recommendations. J Gerontol Nurs. 2009 Mar;35(3):50-7; quiz 58-9. doi: 10.3928/00989134-20090301-03. PMID 19326829
- [Background] Requena C, Lopez Ibor MI, Maestu F, Campo P, Lopez Ibor JJ, Ortiz T. Effects of cholinergic drugs and cognitive training on dementia. Dement Geriatr Cogn Disord. 2004;18(1):50-4. doi: 10.1159/000077735. Epub 2004 Apr 6. PMID 15084794
- [Background] Requena C, Maestu F, Campo P, Fernandez A, Ortiz T. Effects of cholinergic drugs and cognitive training on dementia: 2-year follow-up. Dement Geriatr Cogn Disord. 2006;22(4):339-45. doi: 10.1159/000095600. Epub 2006 Sep 4. PMID 16954689
- [Background] Finn M, McDonald S. A single case study of computerised cognitive training for older persons with mild cognitive impairment. NeuroRehabilitation. 2014 Jan 1;35(2):261-70. doi: 10.3233/NRE-141121. PMID 24990031
- [Background] Sitzer DI, Twamley EW, Jeste DV. Cognitive training in Alzheimer's disease: a meta-analysis of the literature. Acta Psychiatr Scand. 2006 Aug;114(2):75-90. doi: 10.1111/j.1600-0447.2006.00789.x. PMID 16836595
- [Background] Des Roches CA, Balachandran I, Ascenso EM, Tripodis Y, Kiran S. Effectiveness of an impairment-based individualized rehabilitation program using an iPad-based software platform. Front Hum Neurosci. 2015 Jan 5;8:1015. doi: 10.3389/fnhum.2014.01015. eCollection 2014. PMID 25601831
- [Derived] Marin A, DeCaro R, Schiloski K, Elshaar A, Dwyer B, Vives-Rodriguez A, Palumbo R, Turk K, Budson A. Home-Based Electronic Cognitive Therapy in Patients With Alzheimer Disease: Feasibility Randomized Controlled Trial. JMIR Form Res. 2022 Sep 12;6(9):e34450. doi: 10.2196/34450. PMID 36094804